CLINICAL TRIAL: NCT05021991
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose Range Finding Clinical Trial to Evaluate the Efficacy, Tolerability, and Safety of PRAX-944 in the Treatment of Adults With Essential Tremor
Brief Title: A Clinical Trial of 2 Doses of PRAX-944 in Participants With Essential Tremor
Acronym: Essential1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAX-944-222
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Essential Tremor
Keywords: Movement Disorder; Benign Essential Tremor; Familial Tremor; Hereditary Essential Tremor; Movement Disorder Agents; Calcium Channels, T-type
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen 1 (Experimental): Double-blind Part: Oral dosing, once daily in the morning with titration over 56 days to 100 mg PRAX-944: 7 days of 5 mg, 7 days of 10 mg, 7 days of 20 mg, 7 days of 40 mg, 7 days of 60 mg, 7 days of 80 mg, 14 days of 100 mg
  Extension Part: Double-blind Lead-in: Oral dosing, once daily in the morning over 43 days: 100 mg PRAX-944
  Extension Part: Open-label Flexible PRAX-944 Dosing: Oral dosing, once daily in the morning of 20 mg to 100 mg PRAX-944 for 469 days
  Crossover Part: Following double-blind lead-in/open-label: 1:1 randomization to placebo or stable dose of PRAX-944 for 21 days followed by cross-over to either placebo or PRAX-944 oral dosing, once daily in the morning with titration over 7 days (3 days at 20 mg, 4 days at 40 mg) to 60 mg (14 days) before returning to open-label part.
  Interventions: Drug: 100 mg PRAX-944; Drug: 60 mg PRAX-944; Drug: Placebo; Drug: Flexibly dosed 20 mg to 100 mg PRAX-944
- Regimen 2 (Experimental): Double-blind Part: Oral dosing, once daily in the morning with titration over 56 days to 60 mg PRAX-944: 7 days of 5 mg, 7 days of 10 mg, 7 days of 20 mg, 7 days of 40 mg, 28 days of 60 mg
  Extension Part: Double-blind Lead-in: Oral dosing, once daily in the morning with titration over 43 days to 100 mg PRAX-944: 7 days of 80 mg, 36 days of 100 mg
  Extension Part: Open-label Flexible PRAX-944 Dosing: Oral dosing, once daily in the morning of 20 mg to 100 mg PRAX-944 for 469 days
  Crossover Part: Following double-blind lead-in/open-label: 1:1 randomization to placebo or stable dose of PRAX-944 for 21 days followed by cross-over to either placebo or PRAX-944 oral dosing, once daily in the morning with titration over 7 days (3 days at 20 mg, 4 days at 40 mg) to 60 mg (14 days) before returning to open-label part.
  Interventions: Drug: 100 mg PRAX-944; Drug: 60 mg PRAX-944; Drug: Placebo; Drug: Flexibly dosed 20 mg to 100 mg PRAX-944
- Regimen 3 (Placebo Comparator): Double-blind Part: Oral dosing, once daily in the morning: 56 days of placebo
  Extension Part: Double-blind Lead-in: Oral dosing, once daily in the morning with titration over 43 days to 100 mg PRAX-944: 7 days of 5 mg, 7 days of 10 mg, 7 days of 20 mg, 7 days of 40 mg, 7 days of 60 mg, 7 days of 80 mg, 14 days of 100 mg
  Extension Part: Open-label Flexible PRAX-944 Dosing: Oral dosing, once daily in the morning of 20 mg to 100 mg PRAX-944 for 469 days
  Crossover Part: Following double-blind lead-in/open-label: 1:1 randomization to placebo or stable dose of PRAX-944 for 21 days followed by cross-over to either placebo or PRAX-944 oral dosing, once daily in the morning with titration over 7 days (3 days at 20 mg, 4 days at 40 mg) to 60 mg (14 days) before returning to open-label part.
  Interventions: Drug: 100 mg PRAX-944; Drug: 60 mg PRAX-944; Drug: Placebo; Drug: Flexibly dosed 20 mg to 100 mg PRAX-944

INTERVENTIONS:
Drug: 100 mg PRAX-944 — Once daily oral treatment with titration
Drug: 60 mg PRAX-944 — Once daily oral treatment with titration
Drug: Placebo — Once daily oral treatment
Drug: Flexibly dosed 20 mg to 100 mg PRAX-944 — Once daily oral treatment

SUMMARY:
This multi-center, randomized, double-blinded, placebo-controlled, dose-range-finding clinical trial (with an optional Extension comprised of an Extension Double-blind (DB) Lead in Period followed by an Extension Open-label (OL) Period) that will assess the efficacy, safety, and tolerability of PRAX 944 in participants aged 18 years or older who have a diagnosis of Essential Tremor (ET) and have had symptoms for at least 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ET, including: (a) tremor syndrome of bilateral upper limb action tremor, (b) at least 3 years in duration, (c) with or without tremor in other locations (eg, head, voice, or lower limbs), (d) If the symptoms and signs are judged by the investigator to be due to the diagnosis of ET, it is acceptable for them to also have one or more of the following ET plus signs: (i) mild dystonic posturing, (ii) mild rest tremor in the setting of advanced ET and in the absence of other features of Parkinsonism, (iii) intention tremor, (iv) mild increase in tandem gait difficulty.
2. Participant has moderate to severe functional impairment due to tremor as determined by the TETRAS and CGI-S.
3. If currently receiving any medication for ET, is on a stable dose of any of these medications for ET for 1 month prior to Screening and is willing to maintain stable doses throughout the trial. If receiving primidone for ET, is willing and able to discontinue 14 days prior to Day 1.
4. Body mass index (BMI) between 18 and 40 kg/m² (inclusive).

Exclusion Criteria:

1. Sporadically using a benzodiazepine, sleep medication, or anxiolytic that would confound the assessment of tremor.
2. Trauma to the nervous system within 3 months preceding the onset of tremor.
3. History or clinical evidence of other medical, neurological, or psychiatric condition that may explain or cause tremor, including but not limited to Parkinson's disease, Huntington's disease, Alzheimer's disease, cerebellar disease (including spinocerebellar ataxias), primary dystonia, Fragile X Tremor/Ataxia syndrome or family history of Fragile X syndrome, traumatic brain injury, psychogenic tremor, alcohol or benzodiazepine abuse or withdrawal, multiple sclerosis, polyneuropathy, and endocrine states such as hyperthyroidism or unstable treatment of hypothyroidism or medication, food, or supplement induced movement disorders (eg, tremor related to beta agonists or caffeine), or other medical, neurological, or psychiatric conditions that may explain or cause tremor
4. Prior magnetic resonance-guided focused ultrasound or surgical intervention for ET such as deep brain stimulation or thalamotomy.
5. Botulinum toxin injection for ET in the 6 months prior to Baseline.
6. Cala trio health device for ET in the 14 days prior to Baseline and throughout the study.
7. History of substance use disorder consistent with Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria. Participants with a previous diagnosis of substance use disorder who have been in remission for at least 2 years can participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 56 on the modified ADL | 56 days
  The modified ADL is a composite sum of items 1 to 11 of the TETRAS-ADL subscale and items 6 and 7 on the TETRAS-PS. The impact to each function is rated on a 5-point Likert scale from 0 to 4. Before calculating the total score, a scoring adjustment is applied to each item score. The modified ADL score is calculated as the sum of all 13 items (with scoring adjustments) and ranges from 0 to 42 where larger values represent increased direct tremor impact to activities of daily living.

SECONDARY OUTCOMES:
Change from baseline to Day 56 on the Clinical Global Impression-Severity (CGI-S) | 56 days
  The CGI-S assesses the clinician's impression of the participant's current illness state. The clinician should use his/her total clinical experience with this patient population and rate the current severity of the participant's ET on a 7-point scale from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Clinical Global Impression-Improvement (CGI-I) score at Day 56 | 56 days
  The CGI-I assesses the participant's improvement (or worsening). The clinician is required to assess the participant's condition relative to pre-treatment on a 7-point scale from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement/worsening is drug-related or not.
Change from baseline to Day 56 on the TETRAS-ADL score | 56 days
  The TETRAS-ADL subscale is a 12-item assessment of typical daily activities that are impacted by tremor. Activities are assessed in the following functional domains: speaking, feeding, drinking, personal hygiene, dressing, writing, and social activity. The impact to each function is rated on a 5-point Likert scale from 0 to 4. The ADL subscale score is calculated as the sum of all 12 items and ranges from 0 to 48 where larger values represent increased direct tremor impact to activities of daily living.
Change from baseline to Day 56 on the TETRAS-Performance Subscale (PS) total score | 56 days
  There are 9 items covering different body regions in the Performance Subscale. Each Performance Subscale item is rated on a scale of 0 to 4, with higher scores indicating higher tremor severity. Item 4 of the Performance Subscale is the upper limb item. It is comprised of 6 sub-items (4a, 4b, and 4c assessed for both the right and left upper limbs). The Performance subscale score is calculated as the sum of all 9 items and ranges from 0 to 64 where larger values represent higher tremor severity.
Change from baseline to Day 56 on the TETRAS-upper limb (UL) score (TETRAS-PS item 4) | 56 days
  Item 4 of the Performance subscale is the upper limb item. It is comprised of 6 sub-items (4a, 4b, and 4c assessed for both the right and left upper limbs). Each sub-item is rated on a scale from 0 to 4, with higher scores indicating higher tremor amplitude of the upper limb. The upper limb total score is the sum of these 6 sub-items and ranges from 0 to 24 where larger values represent higher tremor severity.
Change from baseline to Day 56 on the TETRAS-combined upper limb (CUL) score (TETRAS-PS sum of items 4, 6, 7, and 8) | 56 days
  The combined upper limb score is the sum of the 6 sub-item scores of the upper limb item and the handwriting and spirals scores. The combined upper limb score ranges from 0 to 32 where larger values represent higher tremor severity.
Patient Global Impression-Change (PGI-C) score at Day 56 | 56 days
  The PGI-C assesses the participant's change in condition. The participant is required to assess their condition relative to Baseline (Pre-dose on Day 1) on a 7-point scale from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the participant believes the change is drug-related or not.
Change from baseline to Days 14, 28, and 42 on the modified ADL | Up to 42 days
  The modified ADL is a composite sum of items 1 to 11 of the TETRAS-ADL subscale and items 6 and 7 on the TETRAS-PS. The impact to each function is rated on a 5-point Likert scale from 0 to 4. Before calculating the total score, a scoring adjustment is applied to each item score. The modified ADL score is calculated as the sum of all 13 items (with scoring adjustments) and ranges from 0 to 42 where larger values represent increased direct tremor impact to activities of daily living.
Change from baseline to Days 14, 28, and 42 on the CGI-S | Up to 42 days
  The CGI-S assesses the clinician's impression of the participant's current illness state. The clinician should use his/her total clinical experience with this patient population and rate the current severity of the participant's ET on a 7-point scale from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Change from baseline to Days 14, 28, and 42 on the TETRAS-ADL total score | Up to 42 days
  The TETRAS-ADL subscale is a 12-item assessment of typical daily activities that are impacted by tremor. Activities are assessed in the following functional domains: speaking, feeding, drinking, personal hygiene, dressing, writing, and social activity. The impact to each function is rated on a 5-point Likert scale from 0 to 4. The ADL subscale score is calculated as the sum of all 12 items and ranges from 0 to 48 where larger values represent increased direct tremor impact to activities of daily living.
Change from baseline to Days 14, 28, and 42 on the TETRAS-UL score | Up to 42 days
  Item 4 of the Performance subscale is the upper limb item. It is comprised of 6 sub-items (4a, 4b, and 4c assessed for both the right and left upper limbs). Each sub-item is rated on a scale from 0 to 4, with higher scores indicating higher tremor amplitude of the upper limb. The upper limb total score is the sum of these 6 sub-items and ranges from 0 to 24 where larger values represent higher tremor severity.
Change from baseline to Days 14, 28, and 42 on the TETRAS-CUL score | Up to 42 days
  The combined upper limb score is the sum of the 6 sub-item scores of the upper limb item and the handwriting and spirals scores. The combined upper limb score ranges from 0 to 32 where larger values represent higher tremor severity.
CGI-I scores at Days 14, 28, and 42 | Up to 42 days
  The CGI-I assesses the participant's improvement (or worsening). The clinician is required to assess the participant's condition relative to pre-treatment on a 7-point scale from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the rater believes the improvement/worsening is drug-related or not.
PGI-C scores at Days 14, 28, and 42 | Up to 42 days
  The PGI-C assesses the participant's improvement (or worsening). The participant is required to assess their condition relative to Baseline (Pre-dose on Day 1) on a 7-point scale from 1 (very much improved) to 7 (very much worse). In all cases, the assessment should be made independent of whether the participant believes the improvement/worsening is drug-related or not.
Change from baseline to Day 42 on the TETRAS-PS total score | 42 days
  There are 9 items covering different body regions in the Performance Subscale. Each Performance Subscale item is rated on a scale of 0 to 4, with higher scores indicating higher tremor severity. Item 4 of the Performance Subscale is the upper limb item. It is comprised of 6 sub-items (4a, 4b, and 4c assessed for both the right and left upper limbs). The Performance subscale score is calculated as the sum of all 9 items and ranges from 0 to 64.
Number of participants with Adverse Events (AE) | Up to 56 days
  The number of participants with Adverse Events (AE) will be reported by preferred term.

CONTACTS AND LOCATIONS:
Overall Officials: Director, Clinical Development, Study Director — Praxis Precision Medicines
Locations (38):
- United States (34):
  - Praxis Research Site, Birmingham, Alabama
  - Praxis Research Site, Little Rock, Arkansas
  - Praxis Research Site, San Diego, California
  - Praxis Research Site, Santa Monica, California
  - Praxis Research Site, Torrance, California
  - Praxis Research Site, Aurora, Colorado
  - Praxis Research Site, Boca Raton, Florida
  - Praxis Research Site, Gainesville, Florida
  - Praxis Research Site, Jacksonville, Florida
  - Praxis Research Site, Port Charlotte, Florida
  - Praxis Research Site, St. Petersburg, Florida
  - Praxis Research Site, Tampa, Florida
  - Praxis Research Site, West Palm Beach, Florida
  - Praxis Research Site, Chicago, Illinois
  - Praxis Research Site, Kansas City, Kansas
  - Praxis Research Site, Louisville, Kentucky
  - Praxis Research Site, Rockville, Maryland
  - Praxis Research Site, Boston, Massachusetts
  - Praxis Research Site, Burlington, Massachusetts
  - Praxis Research Site, Farmington Hills, Michigan
  - Praxis Research Site, Golden Valley, Minnesota
  - Praxis Research Site, Las Vegas, Nevada
  - Praxis Research Site, New York, New York
  - Praxis Research Site, Cincinnati, Ohio
  - Praxis Research Site, Philadelphia, Pennsylvania
  - Praxis Research Site, Georgetown, Texas
  - Praxis Research Site, Houston, Texas
  - Praxis Research Site, Round Rock, Texas
  - Praxis Research Site, Burlington, Vermont
  - Praxis Research Site, Alexandria, Virginia
  - Praxis Research Site, Virginia Beach, Virginia
  - Praxis Research Site, Kirkland, Washington
  - Praxis Research Site, Spokane, Washington
  - Praxis Research Site, Milwaukee, Wisconsin
- Canada (4):
  - Praxis Research Site, Vancouver, British Columbia
  - Praxis Research Site, Halifax, Nova Scotia
  - Praxis Research Site, Toronto, Ontario
  - Praxis Research Site, Montreal, Quebec